CLINICAL TRIAL: NCT02008019
Title: A Randomized Prospective, Multicentric, Open Label, Phase II Study Aiming to Evaluate the Efficacity and Safety of EVEROLIMUS as Neo-adjuvant Therapy in Patients With Primary or Relapsed Chondrosarcomas
Brief Title: A Phase II Study of EVEROLIMUS in Patients With Primary or Relapsed Chondrosarcomas
Acronym: CHONRAD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was suspended since july 27th 2016 because of unavailability of Everolimus
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHONRAD
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Chondrosarcoma
Keywords: Chondrosarcoma; Neoadjuvant therapy; Phase II; Everolimus; Success Rate; Progression Free Survival; Overall Survival; Safety; Quality of Life; Molecular study (ancillary study)
MeSH Terms: conditions — Chondrosarcoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No treatment (No Intervention): No Everolimus treatment before surgery
- Everolimus 2,5 mg/day (Experimental): Everolimus treatment at 2,5 mg/day for 30 days
  Interventions: Drug: Everolimus 2.5 mg/day
- Everolimus 10 mg/day (Experimental): Everolimus treatment at 10 mg/day for 30 days
  Interventions: Drug: Everolimus 10 mg/day

INTERVENTIONS:
Drug: Everolimus 2.5 mg/day — Comparison between 2,5 mg/day of Everolimus per os to 10 mg/day, or to no treatment, taken during 30 days before chondrosarcoma surgery
  Other Names: Afinitor; Votubia; RAD-001
  Arms: Everolimus 2,5 mg/day
Drug: Everolimus 10 mg/day — Comparison between 10 mg/day of Everolimus per os to 2.5 mg/day, or to no treatment taken during 30 days before chondrosarcoma surgery
  Other Names: Afinitor; Votubia; RAD-001
  Arms: Everolimus 10 mg/day

SUMMARY:
The mainstay of chondrosarcoma treatment is a wide surgical resection. Unfortunately, this is a rare occurrence, and patients with incomplete resection have very poor therapeutic options. In this context, it becomes important to find new therapeutic strategies to slow down tumor progression and to reduce tumor size before resection.

Pre-clinical and clinical data suggest that EVEROLIMUS should be efficient as adjuvant and neo-adjuvant therapy in chondrosarcoma.

Then, investigators propose a phase II, randomized, open label study compounded by 3 arms (1:1:1) to assess efficiency of EVEROLIMUS as neo-adjuvant therapy in patients with primary or relapsed chondrosarcomas :

ARM 1 = No treatment; ARM 2 = 2,5 mg Everolimus/day; ARM 3 = 10 mg Everolimus/day.

The treatments will be taken for 4 weeks before surgery, apart from any premature withdrawn

DETAILED DESCRIPTION:
Chondrosarcomas (CHS) represent 25% of bone sarcomas and are the second most frequent primary malignant type of bone tumor. No effective systemic treatment has been identified in advanced or adjuvant phases for CHS. As CHS are relatively resistant to chemo- and radiotherapy, surgery remains the primary treatment of this tumor type. The aim of tumor resection is to obtain complete removal of the malignant lesion with adequate margins taking into account tumor control and functional reconstruction. However, considering the particular localizations of CHS, a wide resection (i.e. R0 clear margins) is rarely achieved. Unfortunately, therapeutic options are limited for patients with incomplete resection. In this context, new therapeutic strategies are needed to slow down tumor progression and to reduce tumor size before surgery.

Increasing knowledge of the signal transduction pathways involved in oncogenesis has led to speculation that components of signalling pathways could be envisaged as novel targets for cancer therapy. Mammalian Target of Rapamycin (mTOR), which lies downstream of the Phosphatidylinositol 3-kinase/B kinase protein (PI3K/Akt) pathway, plays a central role in the regulation of cancer cell growth, suggesting that mTOR could be an attractive target for anti-cancer therapy. The PI3K-Akt-mTOR signaling pathway is intimately implicated in sarcoma development and progression. Indeed, mutations and/ or overexpression of one or several components of the PI3K-Akt-mTOR pathway are often observed in sarcoma. These alterations, located both upstream and downstream of mTOR, lead to dysregulation of the mTOR pathway. mTOR inhibitor evaluation as anticancer agents has began with rapamycin analogues (called rapalogs). Currently, mTOR inhibitors under clinical development include temsirolimus (CCI-779, Torisel®, Wyeth Pharmaceuticals), everolimus (RAD001, Afinitor®, Novartis Pharmaceuticals), and ridaforolimus (AP23573, ARIAD Pharmaceuticals). mTOR inhibitors were found to be efficient in various preclinical cancer models, for example in a preclinical mouse model of follicular thyroid cancer, everolimus induced a significant decrease in proliferation of cancer cells.

Two sets of recent data suggest that inhibition of mTOR pathway could be an effective systemic treatment for chondrosarcoma. The first one is a case report describing an impressive tumor response in a patient with myxoid chondrosarcoma treated by rapamycin in combination with cyclophosphamide. The second one concerns nonclinical data generated by our institution. Using an orthotopic rat chondrosarcoma model, we have shown that monotherapy with everolimus inhibits chondrosarcoma proliferation as evaluated by Ki67 expression and significantly reduced tumor volume. Importantly, when given in a "pseudo-adjuvant" setting following R1 resection of the implanted tumor, everolimus significantly delayed tumor recurrence. These preclinical data provide a strong rationale to evaluate the therapeutic potential of everolimus in both the neo-adjuvant and adjuvant settings in patients with chondrosarcoma.

In this context, the proposal of the investigators is to perform a multicenter, randomized, Phase II study in patients with a primary or relapsed chondrosarcoma in neo-adjuvant setting

ELIGIBILITY:
INCLUSION CRITERIA :

* Male or Female ≥ 18 years
* Histopathologically confirmed diagnosis of primary or relapsed conventional CHS of the bone (with or without metastases), CHS of any size on MRI if relapse OR size ≥ 10 cm on MRI at diagnosis OR CHS < 10 cm if R0 resection with adequate margins is not feasible at 1st examination (localization, tumor infiltration within surrounding tissues).
* Patient with life expectancy > 6 months
* Planned surgery between D32- D40 after inclusion
* Performance status of Eastern Cooperative Oncology Group (ECOG) ≤ 2
* No contra-indication to Everolimus as per Summary of Product Characteristics (SPC)
* Adequate bone marrow, liver and renal functions including the following:

  * Hemoglobin > 9 g/dL
  * Neutrophil count ≥ 1500 x 109/L
  * Platelets ≥ 100 x 109/L
  * Total bilirubin ≤ 1,5x upper limit of normal (ULN)
  * Serum Glutamate Oxaloacetate Transaminase (SGOT) and Serum Glutamate Pyruvate Transaminase (SGPT) ≤ 3 x ULN
  * Alkaline Phosphatase ≤ 2,5 x ULN
  * Serum creatinine < 110 µmol/L or creatinine clearance > 55 ml/min (estimated by Cockcroft Formula)
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Ability to understand and willingness to sign a written informed consent
* In accordance with French Regulatory Authorities: Patients with French Social Security in compliance with the French law relating to biomedical research (Huriet Law 88-1128 and related decrees)
* Women of child-bearing potential and men must agree to use adequate double contraception prior to study entry, for the duration of study participation and 30 days after the last study drug intake.

EXCLUSION CRITERIA :

* Mesenchymal, dedifferentiated, clear cell subtype chondrosarcoma, and soft tissues chondrosarcoma
* Tumor tissue sample not available for pathological review/or correlative studies
* Patients may not be receiving any other investigational agents
* Prior treatment with mTOR inhibitors
* Symptomatic congestive heart failure of New York heart Association Class III or IV
* Uncontrolled diabetes as defined by fasting serum glucose >160 mg/dl or 8.9 mmol/l
* Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* Chemotherapy within the last 4 weeks before inclusion; radiotherapy, or any other investigational agent within 14 days or 5 half-lives, whichever is longer prior to the first dose of study drug
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Impaired cardiac function or clinically significant cardiac diseases, or liver, respiratory or hepatic disease
* Known diagnosis of HIV infection
* Patient with ongoing toxicity Grade ≥ 2 according to the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0
* Pregnant or breast feeding women (a pregnancy test will be performed within 7 days before inclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2014-08-14 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Success Rate obtained per arm | 4 weeks after inclusion
  A success is defined as a variation (decrease) of Ki67 expression > 10% during treatment

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | At time of progression in the course of the 3 years follow up after randomization
  PFS = Time from randomization until the date of event defined as the first documented progression or death due to any cause. Patients without any progression at the end of the 3 years follow up will be censured at this date.
Safety | In the course of the 3 years after randomization
  Based on the frequency of Adverse Events according to common toxicity criteria (CTC V4.0), taking to account post operative complications and functional outcomes
Overall Survival | At time of death if occuring during the 3 years of follow up after randomization
  Patients who are alive at the end of the 3 years follow up will be censured at this date.
Quality of Life | From randomization to the end of the 3 years follow up
  Data collected from a questionnaire at inclusion, surgery, 3th month, 6th month, 12th month, 24th month and 36th month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, Professor, Principal Investigator — Centre Léon Bérard, Lyon; François Gouin, Professor, Principal Investigator — Centre Hospitalier Universitaire de Nantes, Hôtel Dieu
Locations (12):
- France (12):
  - Institut Bergonié, Bordeaux, Gironde
  - Institut Claudius Regaud, Toulouse, Haute Garonne
  - Centre Hospitalier Universitaire de Limoges, Hôpital Dupuytren, Limoges, Haute Vienne
  - Institut Régional du Cancer de Montpellier, Montpellier, Hérault
  - Centre Hospitalier Régional Universitaire de Tours, Hôpital Trousseau, Tours, Indre et Loire
  - Centre Hospitalier Universitaire de Nantes, Hôtel Dieu, Nantes, Loire Atlantique
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain, Loire Atlantique
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, Meurthe et Moselle
  - Centre Oscar Lambret, Lille, Nord
  - CHRU de Lille - Hôpital Roger Salengro, Lille, Nord
  - Centre Léon Bérard, Lyon, Rhône
  - Institut Gustave Roussy, Villejuif, Val de Marne

REFERENCES:
- [Background] Lichtenstein L, Jaffe HL. Chondrosarcoma of Bone. Am J Pathol. 1943 Jul;19(4):553-89. No abstract available. PMID 19970709
- [Background] Dahlin DC, Unni KK Bone tumors: general aspects and data on 8542 cases. Fourth ed. Sprinfield, Illinois: Charles C Thomas,1986.
- [Background] Enneking WF. Musculoskeletal tumor surgery. Vol 2. New York, Churchill Livingstone, 1983: 875-997.
- [Background] O'NEAL LW, ACKERMAN LV. Chondrosarcoma of bone. Cancer. 1952 May;5(3):551-77. doi: 10.1002/1097-0142(195205)5:33.0.co;2-z. No abstract available. PMID 14925925
- [Background] Fiorenza F, Abudu A, Grimer RJ, Carter SR, Tillman RM, Ayoub K, Mangham DC, Davies AM. Risk factors for survival and local control in chondrosarcoma of bone. J Bone Joint Surg Br. 2002 Jan;84(1):93-9. doi: 10.1302/0301-620x.84b1.11942. PMID 11837841
- [Background] Lee FY, Mankin HJ, Fondren G, Gebhardt MC, Springfield DS, Rosenberg AE, Jennings LC. Chondrosarcoma of bone: an assessment of outcome. J Bone Joint Surg Am. 1999 Mar;81(3):326-38. doi: 10.2106/00004623-199903000-00004. PMID 10199270
- [Background] Pritchard DJ, Lunke RJ, Taylor WF, Dahlin DC, Medley BE. Chondrosarcoma: a clinicopathologic and statistical analysis. Cancer. 1980 Jan 1;45(1):149-57. doi: 10.1002/1097-0142(19800101)45:13.0.co;2-a. PMID 7350999
- [Background] Gitelis S, Bertoni F, Picci P, Campanacci M. Chondrosarcoma of bone. The experience at the Istituto Ortopedico Rizzoli. J Bone Joint Surg Am. 1981 Oct;63(8):1248-57. PMID 7287795
- [Background] Evans HL, Ayala AG, Romsdahl MM. Prognostic factors in chondrosarcoma of bone: a clinicopathologic analysis with emphasis on histologic grading. Cancer. 1977 Aug;40(2):818-31. doi: 10.1002/1097-0142(197708)40:23.0.co;2-b. No abstract available. PMID 890662
- [Background] Pring ME, Weber KL, Unni KK, Sim FH. Chondrosarcoma of the pelvis. A review of sixty-four cases. J Bone Joint Surg Am. 2001 Nov;83(11):1630-42. PMID 11701784
- [Background] Miser JS, Pappo AS, Triche TJ et al. In: Pizzo PA, Poplack DG, eds. Principles and Practice of Pediatric Oncology. Other soft tissue sarcomas of childhood. Philadelphia, PA: Lippincott Williams & Wilkins, 2002:1017-1050.
- [Background] Marina N, Gebhardt M, Teot L, Gorlick R. Biology and therapeutic advances for pediatric osteosarcoma. Oncologist. 2004;9(4):422-41. doi: 10.1634/theoncologist.9-4-422. PMID 15266096
- [Background] Fingar DC, Blenis J. Target of rapamycin (TOR): an integrator of nutrient and growth factor signals and coordinator of cell growth and cell cycle progression. Oncogene. 2004 Apr 19;23(18):3151-71. doi: 10.1038/sj.onc.1207542. PMID 15094765
- [Background] Hay N, Sonenberg N. Upstream and downstream of mTOR. Genes Dev. 2004 Aug 15;18(16):1926-45. doi: 10.1101/gad.1212704. PMID 15314020
- [Background] Faivre S, Kroemer G, Raymond E. Current development of mTOR inhibitors as anticancer agents. Nat Rev Drug Discov. 2006 Aug;5(8):671-88. doi: 10.1038/nrd2062. PMID 16883305
- [Background] Wan X, Mendoza A, Khanna C, Helman LJ. Rapamycin inhibits ezrin-mediated metastatic behavior in a murine model of osteosarcoma. Cancer Res. 2005 Mar 15;65(6):2406-11. doi: 10.1158/0008-5472.CAN-04-3135. PMID 15781656
- [Background] Raymond E, Alexandre J, Faivre S, Vera K, Materman E, Boni J, Leister C, Korth-Bradley J, Hanauske A, Armand JP. Safety and pharmacokinetics of escalated doses of weekly intravenous infusion of CCI-779, a novel mTOR inhibitor, in patients with cancer. J Clin Oncol. 2004 Jun 15;22(12):2336-47. doi: 10.1200/JCO.2004.08.116. Epub 2004 May 10. PMID 15136596
- [Background] Huang S, Houghton PJ. Inhibitors of mammalian target of rapamycin as novel antitumor agents: from bench to clinic. Curr Opin Investig Drugs. 2002 Feb;3(2):295-304. PMID 12020063
- [Background] Galanis E, Buckner JC, Maurer MJ, Kreisberg JI, Ballman K, Boni J, Peralba JM, Jenkins RB, Dakhil SR, Morton RF, Jaeckle KA, Scheithauer BW, Dancey J, Hidalgo M, Walsh DJ; North Central Cancer Treatment Group. Phase II trial of temsirolimus (CCI-779) in recurrent glioblastoma multiforme: a North Central Cancer Treatment Group Study. J Clin Oncol. 2005 Aug 10;23(23):5294-304. doi: 10.1200/JCO.2005.23.622. Epub 2005 Jul 5. PMID 15998902
- [Background] O'Donnell A, Faivre S, Judson I et al. A phase I study of the oral mTOR inhibitors RAD001 as monotherapy to identify the optimal biologically effective dose using toxicity, pharmacokinetic (PK) and pharmacodynamic (PD) endpoints in patients with solid tumors. Proc Am Soc Clin Oncol 2003;22:803a
- [Background] Dudkin L, Dilling MB, Cheshire PJ, Harwood FC, Hollingshead M, Arbuck SG, Travis R, Sausville EA, Houghton PJ. Biochemical correlates of mTOR inhibition by the rapamycin ester CCI-779 and tumor growth inhibition. Clin Cancer Res. 2001 Jun;7(6):1758-64. PMID 11410517
- [Background] Hidalgo M, Rowinsky EK. The rapamycin-sensitive signal transduction pathway as a target for cancer therapy. Oncogene. 2000 Dec 27;19(56):6680-6. doi: 10.1038/sj.onc.1204091. PMID 11426655
- [Background] Amornphimoltham P, Patel V, Sodhi A, Nikitakis NG, Sauk JJ, Sausville EA, Molinolo AA, Gutkind JS. Mammalian target of rapamycin, a molecular target in squamous cell carcinomas of the head and neck. Cancer Res. 2005 Nov 1;65(21):9953-61. doi: 10.1158/0008-5472.CAN-05-0921. PMID 16267020
- [Background] Guigon CJ, Fozzatti L, Lu C, Willingham MC, Cheng SY. Inhibition of mTORC1 signaling reduces tumor growth but does not prevent cancer progression in a mouse model of thyroid cancer. Carcinogenesis. 2010 Jul;31(7):1284-91. doi: 10.1093/carcin/bgq059. Epub 2010 Mar 18. PMID 20299527
- [Background] Meric-Bernstam F, Gonzalez-Angulo AM. Targeting the mTOR signaling network for cancer therapy. J Clin Oncol. 2009 May 1;27(13):2278-87. doi: 10.1200/JCO.2008.20.0766. Epub 2009 Mar 30. PMID 19332717
- [Background] MacKenzie AR, von Mehren M. Mechanisms of mammalian target of rapamycin inhibition in sarcoma: present and future. Expert Rev Anticancer Ther. 2007 Aug;7(8):1145-54. doi: 10.1586/14737140.7.8.1145. PMID 18028023
- [Background] Mita M, Sankhala K, Abdel-Karim I, Mita A, Giles F. Deforolimus (AP23573) a novel mTOR inhibitor in clinical development. Expert Opin Investig Drugs. 2008 Dec;17(12):1947-54. doi: 10.1517/13543780802556485. PMID 19012509
- [Background] Mahalingam D, Mita A, Sankhala K, Swords R, Kelly K, Giles F, Mita MM. Targeting sarcomas: novel biological agents and future perspectives. Curr Drug Targets. 2009 Oct;10(10):937-49. doi: 10.2174/138945009789577990. PMID 19860642
- [Background] Merimsky O, Bernstein-Molho R, Sagi-Eisenberg R. Targeting the mammalian target of rapamycin in myxoid chondrosarcoma. Anticancer Drugs. 2008 Nov;19(10):1019-21. doi: 10.1097/CAD.0b013e328312c0e5. PMID 18827568
- [Background] Enneking WF, Dunham W, Gebhardt MC, Malawar M, Pritchard DJ. A system for the functional evaluation of reconstructive procedures after surgical treatment of tumors of the musculoskeletal system. Clin Orthop Relat Res. 1993 Jan;(286):241-6. PMID 8425352